CLINICAL TRIAL: NCT04410094
Title: A Phase 1 Open-Label, Fixed-Sequence Drug-Drug Interaction Study to Evaluate the Effects of Steady-state Itraconazole and Rifampin on the Single-dose Pharmacokinetics of Lazertinib Tablets in Healthy Adult Participants
Brief Title: A Study to Assess the Effects of Itraconazole and Rifampin on Lazertinib in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108799; 73841937NSC1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Healthy
MeSH Terms: interventions — lazertinib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Lazertinib plus Itraconazole (Experimental): Participants will receive a single oral dose of lazertinib tablets in Treatment Period 1 followed by itraconazole capsules orally along with a single oral dose of lazertinib tablet in Treatment Period 2.
  Interventions: Drug: Lazertinib; Drug: Itraconazole
- Cohort 2: Lazertinib plus Rifampin (Experimental): Participants will receive a single oral dose of lazertinib tablets in Treatment Period 1 followed by rifampin capsules orally along with a single oral dose of lazertinib tablet in Treatment Period 2.
  Interventions: Drug: Lazertinib; Drug: Rifampin

INTERVENTIONS:
Drug: Lazertinib — Lazertinib tablets will be administered orally.
  Other Names: JNJ-73841937; YH25448
Drug: Itraconazole — Itraconazole capsules will be administered orally.
  Arms: Cohort 1: Lazertinib plus Itraconazole
Drug: Rifampin — Rifampin capsules will be administered orally.
  Arms: Cohort 2: Lazertinib plus Rifampin

SUMMARY:
The purpose of this study is to evaluate the effects of multiple doses of strong cytochrome P450 (CYP) 3A4 inhibitor itraconazole and strong CYP3A4 inducer rifampin on the single dose pharmacokinetics (PK) of lazertinib in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* A woman must not be of childbearing potential and must have a negative serum beta-human chorionic gonadotropin (Beta HCG) pregnancy test at screening
* Hormone replacement therapy (if applicable) must have been discontinued at least 28 days prior to the first dose of study drug (Cohort 2 only)
* Participants must have a body mass index (BMI) between 18.0 and 32.0 kilogram per meter square (kg/m^2, inclusive (BMI = weight/height^2), and body weight not less than 50 kg at screening
* Participants must be healthy based on physical examination, medical history, and vital signs (pulse and body temperature), performed at screening
* Male participants must agree to use an adequate contraception method

Exclusion Criteria:

* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of infection suspected or confirmed to be related to Coronavirus disease 2019 (COVID-19) within 4 weeks before intake of study drug
* Participant has known allergies, hypersensitivity, or intolerance to lazertinib or its excipients or to itraconazole and rifampin
* Participant has contraindications to the use itraconazole and rifampin per local prescribing information
* Use of any cytochrome P450 (CYP) 3A4 inhibitors or inducers (other than per-protocol itraconazole/rifampin administration) within 4 weeks before the first dose of the study drug is scheduled until completion of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Cohort 1 and 2: Maximum Plasma Concentration (Cmax) of Lazertinib | Predose up to 120 hours post dose
  Cmax is defined as maximum plasma concentration.
Cohort 1 and 2: Area Under the Plasma Concentration-time Curve from Time 0 to 120 Hours (AUC [0-120h]) of Lazertinib | Predose up to 120 hours post dose
  AUC (0-120h) is defined as area under the plasma concentration-time curve from time 0 to 120 hours postdose.
Cohort 1 and 2: Area Under the Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Timepoint (AUC [0-last]) of Lazertinib | Predose up to 120 hours post dose
  AUC (0-last) is defined as area under the plasma concentration-time curve from time 0 to time of last quantifiable timepoint.
Cohort 1 and 2: Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC [0-inf]) of Lazertinib | Predose up to 120 hours post dose
  AUC (0-inf) is defined as area under the plasma concentration-time curve from time 0 to infinity, calculated as the sum of AUC(0-last)+C(last)/ lambda(z), where C(last) is the last observed measurable (non-below limit of quantification) concentration.
Cohort 1 and 2: Percentage of Area Under the Plasma Concentration from time Zero to Infinite time obtained by Extrapolation (%AUC [0-inf],ex) of Lazertinib | Predose up to 120 hours post dose
  %AUC (0-inf),ex is defined as percentage of area under the plasma concentration from time zero to infinite time obtained by extrapolation, calculated as (AUC [0-infinity] minus AUC [0-last]/AUC [0-infinity])*100.

SECONDARY OUTCOMES:
Cohort 1 and Cohort 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 65 days (Cohort 1) and up to 70 days (Cohort 2)
  An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency